CLINICAL TRIAL: NCT04862286
Title: OptIMMize-2: A Phase 3 Multicenter, Single-arm, Open-label Extension Study to Assess the Safety, Tolerability, and Efficacy of Risankizumab in Subjects With Moderate to Severe Plaque Psoriasis Who Have Completed Participation in Study M19-977 (OptIMMize-1)
Brief Title: Study to Evaluate Adverse Events and Change in Disease Activity in Participants Between 6 and 17 Years With Moderate to Severe Plaque Psoriasis Treated With Subcutaneous (SC) Injection of Risankizumab Who Have Completed Participation in Study M19-977
Acronym: OptIMMize-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M19-973; 2022-500408-22-00 (Other: EU CT)
Record Dates: First submitted 2021-04-26; First posted 2021-04-27 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Psoriasis
Keywords: Plaque Psoriasis; Risankizumab; SKYRIZI; ABBV-066; BI 655066; Risankizumab-rzaa
MeSH Terms: conditions — Psoriasis | interventions — risankizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Risankizumab (Experimental): Participants will receive risankizumab subcutaneous (SC) injection every 12 weeks for 204 weeks.
  Interventions: Drug: Risankizumab

INTERVENTIONS:
Drug: Risankizumab — Subcutaneous (SC) injection.
  Other Names: ABBV-066; BI 655066; SKYRIZI; risankizumab-rzaa

SUMMARY:
Psoriasis is a chronic, systemic, inflammatory disease in which skin cells build up and develop thick, red and white scaly patches on the skin. This study evaluates adverse events and change in disease activity with risankizumab in pediatric participants with moderate to severe plaque psoriasis who completed the study M19-977.

Risankizumab is an approved drug for treatment of moderate to severe plaque psoriasis in adults and is being studied in the pediatric population (6 to 17 years). A maximum of 132 participants will be enrolled in the study across approximately 50 sites worldwide.

Participants will receive subcutaneous injection of risankizumab every 12 weeks for 204 weeks and are followed up for safety for 20 weeks after last dose.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

--Participants who have completed participation in study M19-977 and who meet all eligibility criteria for participation in Study M19-973 will be allowed to enroll in study M19-973.

Exclusion Criteria:

--Participants who have developed any discontinuation criteria as defined in Study M19-977.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 132 (Estimated)
Dates: Start 2021-07-24 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | Up to approximately 224 weeks
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either probably related, possibly related, probably not related or not related. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent any of the outcomes listed above.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (41):
- United States (15):
  - UAB Department of Dermatology /ID# 252305, Birmingham, Alabama
  - First OC Dermatology /ID# 226942, Fountain Valley, California
  - Integrative Skin Science and Research /ID# 226108, Sacramento, California
  - University of California San Diego - Rady Children's Hospital San Diego /ID# 252348, San Diego, California
  - Solutions Through Adv Rch /ID# 226104, Jacksonville, Florida
  - Olympian Clinical Research- St. Petersburg /ID# 226106, St. Petersburg, Florida
  - Advanced Clinical Research Institute /ID# 248827, Tampa, Florida
  - University Dermatology and Vein Clinic, LLC /ID# 226100, Darien, Illinois
  - Arlington Dermatology /ID# 226097, Rolling Meadows, Illinois
  - Skin Cancer and Dermatology Institute - Reno /ID# 248828, Reno, Nevada
  - Univ Hosp Cleveland /ID# 248825, Cleveland, Ohio
  - Apex Clinical Research Center /ID# 248830, Mayfield Heights, Ohio
  - Medical University of South Carolina /ID# 248831, Charleston, South Carolina
  - West Virginia University Hospitals /ID# 263438, Morgantown, West Virginia
  - Wisconsin Medical Center /ID# 263437, Milwaukee, Wisconsin
- Canada (2):
  - Karma Clinical Trials /ID# 233985, St. John's, Newfoundland and Labrador
  - Hospital for Sick Children /ID# 233986, Toronto, Ontario
- Germany (6):
  - Fachklinik Bad Bentheim /ID# 243904, Bad Bentheim, Lower Saxony
  - Universitaetsklinikum Bonn /ID# 243910, Bonn, North Rhine-Westphalia
  - Universitaetsklinikum Muenster /ID# 243905, Münster, North Rhine-Westphalia
  - Universitaetsmedizin Mainz /ID# 243907, Mainz, Rhineland-Palatinate
  - Universitaetsklinikum Carl Gustav Carus Dresden /ID# 243908, Dresden, Saxony
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel /ID# 243883, Kiel, Schleswig-Holstein
- Japan (4):
  - Nagoya City University Hospital /ID# 248429, Nagoya, Aichi-ken
  - Mie University Hospital /ID# 263008, Tsu, Mie-ken
  - Kansai Medical University Hirakata Hospital /ID# 252332, Hirakata-shi, Osaka
  - Tokyo Medical University Hospital /ID# 252331, Shinjuku-ku, Tokyo
- Poland (5):
  - High-Med Przychodnia Specjalistyczna /ID# 243846, Warsaw, Masovian Voivodeship
  - Uniwersytecki Szpital Kliniczny im. F. Chopina w Rzeszowie /ID# 243850, Rzeszów, Podkarpackie Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o. /ID# 243849, Gdansk, Pomeranian Voivodeship
  - Dermed Centrum Medyczne Sp. z o.o /ID# 243847, Lodz, Łódź Voivodeship
  - Dermoklinika Medical Center /ID# 243848, Lodz, Łódź Voivodeship
- Spain (5):
  - Hospital Sant Joan de Deu /ID# 241103, Esplugues de Llobregat, Barcelona
  - Hospital General Universitario Gregorio Maranon /ID# 241099, Madrid
  - Hospital Universitario Infanta Leonor /ID# 241100, Madrid
  - Hospital Universitario 12 de Octubre /ID# 241102, Madrid
  - Complejo Hospitalario Universitario de Pontevedra /ID# 241101, Pontevedra
- United Kingdom (4):
  - Royal Devon & Exeter Hospital /ID# 245101, Exeter, Devon
  - Derriford Hospital and the Royal Eye Infirmary /ID# 245104, Plymouth, Devon
  - Dup_Guys and St Thomas NHS Foundation Trust - Guy's Hospital /ID# 245100, London, Greater London
  - Chelsea and Westminster Hospital /ID# 245102, London, Greater London

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com/